CLINICAL TRIAL: NCT02714504
Title: Evaluation of the Efficacy of Anti-mold Azole Prophylaxis in High-risk Hematologic Patients With Baseline Superficial Skin Lesions Positive for Fusarium Spp
Brief Title: Anti-mold Azole in the Prophylaxis for Invasive Fusariosis
Acronym: Fusarproph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Marcio Nucci, Associate Professor, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Fusarium prophylaxis
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-01

CONDITIONS: Fusariosis; Onychomycosis
Keywords: Prophylaxis
MeSH Terms: conditions — Fusariosis; Onychomycosis | interventions — Voriconazole; posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observational (No Intervention): No anti-mold prophylaxis given on the basis of results of baseline presence of skin lesions
- Anti-mold prophylaxis (Experimental): Anti-mold prophylaxis with either voriconazole or posaconazole for patients with baseline skin lesions in the extremities positive for Fusarium spp.
  Interventions: Drug: Voriconazole or posaconazole

INTERVENTIONS:
Drug: Voriconazole or posaconazole — Azole with activity against molds
  Arms: Anti-mold prophylaxis

SUMMARY:
Patients admitted for autologous or allogeneic hematopoietic cell transplantation, induction-remission chemotherapy for acute myeloid leukemia, myelodysplasia or acute lymphoid leukemia, or to receive immunosuppressive therapy for aplastic anemia will be screened with dermatologic examination. In the presence of any skin lesion in the extremities, direct exam and fungal culture will be performed. If these exams indicate the presence of Fusarium species, patients will receive anti-mold azole prophylaxis

DETAILED DESCRIPTION:
Patients admitted for autologous or allogeneic hematopoietic cell transplantation, induction-remission chemotherapy for acute myeloid leukemia, myelodysplasia or acute lymphoid leukemia, or to receive immunosuppressive therapy for aplastic anemia will be screened on admission. Patients may be included more than once, provided that a new treatment is administered and >30 days elapses from one to other admission (episode).

Screening will consist of a thorough physical examination in the extremities. In case of a skin lesion, direct exam and fungal culture will be performed. Nail samples will be obtained by scrapping the nails with a curette, and samples from interdigital areas will be obtained using swabs.

In a first phase no intervention will be performed. In a second phase, if direct exam and /or culture indicate the presence of Fusarium spp., primary antifungal therapy with an anti-mold azole (voriconazole (200 mg BID) or posaconazole (200 mg TID) will be started.

Patients will be followed until discharge. The primary endpoint is invasive fusariosis, comparing the observational period with the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* admission for autologous or allogeneic hematopoietic cell transplantation, induction-remission chemotherapy for acute myeloid leukemia, myelodysplasia or acute lymphoid leukemia, or to receive immunosuppressive therapy for aplastic anemia

Exclusion Criteria:

* prior documentation of invasive fusariosis or allergy to azoles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational | Anti-mold Prophylaxis
Started | 61 | 178
Completed | 61 | 178
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observational | Anti-mold Prophylaxis | Total
Number analyzed (Participants) | 61 | 178 | 239
Age, Continuous [Median (Full Range); unit: years]
  Age | 44 [14 to 66] | 50 [13 to 72] | 48 [13 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 109 | 146
  Male | 24 | 69 | 93

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Develop Invasive Fusariosis Until Neutrophil Recovery
Description: Proportion of patients who develop invasive fusariosis until neutrophil recovery, for an average of 4 weeks
Time Frame: Until neutrophil recovery, for an average of 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Anti-mold Prophylaxis
Number analyzed (Participants) | 61 | 178
Participants | 6 | 8

ADVERSE EVENTS:
Arm/Group | Observational | Anti-mold Prophylaxis
All-Cause Mortality (participants affected / at risk) | 11/61 | 18/178
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/178
Other Adverse Events (participants affected / at risk) | 0/61 | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes